Official title: Impact of exercise on expression of Hsp70 in individuals at risk of peripheral arterial disease.

**NCT ID: Not yet assigned** 

Document's date: June 3, 2019

## **INFORMED CONSENT LETTER**

| Introduction / Objective: |
|---|
| I, (name) |
| Signature:, of (age) years old, am invited to participate in the protocol "Impact of exercise on expression of Hsp70 in individuals a risk of peripheral arterial disease". |
| The objective of the study is to determine the serum expression level of the HSP70 protein in individuals at risk of atherosclerotic peripheral arterial disease, after a moderate exercise intervention. |
| <b>Procedures and potential risks</b> : If I agree to participate in the study, the procedure is as follows: I will be given a survey that includes personal data, I will perform a stress test, declare that I am not aware of having any heart or lung disease, as well as no cardiac facto that prevents me from doing this activity. |
| Two blood samples from my forearm will be taken of me, with a difference of 3 months which have a risk of pain from the puncture with a needle, bruising (collection of blood unde the skin) may even damage some nerve in the area where it is punctured. |
| I will do moderate exercise sessions for 3 months. This exercise program has inherent risks because of my age. In that case I will receive the corresponding medical attention. |
| <b>Benefits</b> : The benefit of my participation in the study will be to receive recommendations or diet, follow-up from internal medicine, as well as recommendations to follow a home. Receive a sheet with the most relevant data of my assessment. Receive exercise sessions for 3 months. |
| <b>Confidentiality</b> : All the information collected about me and the data obtained will be strictly confidential. They will be used only for health purposes. I can request updated information from the responsible researcher during the study. |
| <b>Voluntary Participation / Withdrawal</b> : I can withdraw from the project if I consider is convenient to my interests, even when the responsible researcher does not request it stating my reasons for such decision. There will be no unfavorable consequence for my personal integrity if I do not accept. |
| Place and date: Name and signature of the responsible researcher: Witness: Name: Signature: |